CLINICAL TRIAL: NCT02480439
Title: A Phase 1, Randomized, Open-Label, Single-Dose, 3-Way Crossover Study to Assess the Relative Bioavailability of a TAK-648 Tablet Compared With a TAK-648 Oral Solution, and to Assess the Effect of Food on the Bioavailability of a TAK-648 Tablet in Healthy Participants
Brief Title: A Study to Assess the Relative Bioavailability and to Assess the Effect of Food on the Bioavailability of a TAK-648 Tablet in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TAK-648-1003; U1111-1170-0503 (Registry Identifier: WHO)
Record Dates: First submitted 2015-06-19; First posted 2015-06-24 (Estimated); Results first posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-07

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- TAK-648 Sequence ABC (Experimental): Regimen A TAK-648 0.3 mg, tablet, orally, 30 minutes after a high fat meal, once on Day 1 of Period 1, followed by at least 7 day washout period, followed by Regimen B TAK-648 0.3 mg, tablet, orally, in fasted state, once on Day 1 of Period 2, followed by at least 7 day washout period, followed by Regimen C TAK-648 0.3 mg, solution, orally, in fasted state, once on Day 1 of Period 3.
  Interventions: Drug: TAK-648 Tablet; Drug: TAK-648 Oral Solution
- TAK-648 Sequence BCA (Experimental): Regimen B TAK-648 0.3 mg, tablet, orally, in fasted state, once on Day 1 of Period 1, followed by at least 7 day washout period, followed by Regimen C TAK-648 0.3 mg, solution, orally, in fasted state, once on Day 1 of Period 2, followed by at least 7 day washout period, followed by Regimen A TAK-648 0.3 mg, tablet, orally, 30 minutes after a high fat meal, once on Day 1 of Period 3.
  Interventions: Drug: TAK-648 Tablet; Drug: TAK-648 Oral Solution
- TAK-648 Sequence CAB (Experimental): Regimen C TAK-648 0.3 mg, solution, orally, in fasted state, once on Day 1 of Period 1, followed by at least 7 day washout period, followed by Regimen A TAK-648 0.3 mg, tablet, orally, after a high fat meal, once on Day 1 of Period 2, followed by at least 7 day washout period, followed by Regimen B TAK-648 0.3 mg, tablet, orally, in fasted state, once on Day 1 of Period 3.
  Interventions: Drug: TAK-648 Tablet; Drug: TAK-648 Oral Solution

INTERVENTIONS:
Drug: TAK-648 Tablet — Tak-648 tablet
Drug: TAK-648 Oral Solution — TAK-648 oral solution

SUMMARY:
The purpose of this study is to assess the relative bioavailability of a TAK-648 tablet compared with a TAK-648 oral solution, and to assess the effect of food on the bioavailability of a TAK-648 tablet in healthy participants.

DETAILED DESCRIPTION:
This study will assess the relative Bioavailability (BA) of TAK-648 tablet compared with that of TAK-648 solution and the effect of food on the BA of the TAK-648 tablet.

The study will enroll approximately 24 healthy participants. Participants will be randomly assigned to one of the three treatment sequences:

* TAK-648 tablet in fed state, followed by TAK-648 tablet in fasted state, followed by TAK-648 oral solution in fasted state
* TAK-648 tablet in fasted state, followed by TAK-648 oral solution in fasted state, followed by TAK-648 tablet in fed state
* TAK-648 oral solution in fasted state, TAK-648 tablet in fed state, TAK-648 tablet in fasted state The dosing in a period and the subsequent period will be separated by a minimum 7-day washout interval. Participants will be asked to take single dose of TAK-648 tablet or oral solution on Day 1 of each period.

This single-center trial will be conducted in the United States. Participants will make 4 visits to the clinic including three 4-day periods of confinement to the clinic, and will be contacted by telephone 30 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female aged 18 to 55 years, inclusive, at the time of informed consent and first study medication dose.
2. Weighs at least 50 kilogram (kg) (110 pounds [lbs]) and has a body mass index (BMI) from 18.0 to 30.0 kilogram per square meter (kg/m^2), inclusive at Screening.
3. Has systolic blood pressure greater than (>) 90 and less than or equal to (<=) 150 millimeter of mercury (mmHg) and diastolic blood pressure >60 and <=90 mm Hg at Screening and at Check-in (Day -1) of Period 1. If out of range, may be repeated once for eligibility determination within a maximum of 5 minutes.
4. Has a calculated creatinine clearance >60 milliliter per minute (mL/min) at Screening and Check-in (Day -1) of Period 1.
5. Male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 12 weeks after last dose.
6. Female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent and throughout the duration of the study and for 12 weeks after the last dose.

Exclusion Criteria:

1. Has received any investigational compound within 30 days prior to the first dose of study medication.
2. Has received TAK-648 in a previous clinical study or as a therapeutic agent.
3. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in the conduct of this study (example, spouse, parent, child, sibling) or may consent under duress.
4. Has any significant medical histories or currently uncontrolled clinical conditions, which may render it unsafe for participant to participate in the study, may impact the ability of the participant to participate in the study, or may potentially confound the study results.
5. Has a history of significant gastrointestinal (GI) disorders manifested with persistent, chronic, or intermittent nausea, vomiting, or diarrhea, or has a current or recent (within 6 months) GI disease that would influence the absorption of drugs.
6. Has diagnosis of major depression, bipolar disorder, or anxiety disorders, or has received any medication to treat any psychological disorders within 1 year.
7. Has a risk of suicide according to the investigator's clinical judgment per Columbia-Suicide Severity Rating Scale (C-SSRS) at screening or has made a suicide attempt in the past 6 months prior to screening.
8. Has known hypersensitivity to any component of the formulation of TAK-648, or to a phosphodiesterase type 4 (PDE4) inhibitor (example, roflumilast).
9. Has taken any excluded medication, supplements, or food products during the time periods listed in the Prohibited Medications table.
10. Has abnormal Screening or Check-in (Day -1) of Period 1 laboratory values that suggest a clinically significant underlying disease or participant has the following laboratory abnormalities: Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >2.5* upper limit of normal (ULN).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 23 June 2015 to 02 September 2015.
Pre-assignment Details: Healthy participants were enrolled equally in 1 of 3 treatment sequences that determined the order of the three treatments received: TAK-648 0.3 mg tablet (fed), 0.3 mg tablet (fasted) and 0.3 mg solution (fasted).
Period: Treatment Period 1
Arm/Group | TAK-648 Sequence ABC | TAK-648 Sequence BCA | TAK-648 Sequence CAB
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | TAK-648 Sequence ABC | TAK-648 Sequence BCA | TAK-648 Sequence CAB
Started | 8 | 7 (1 Participant was withdrawn due to an Adverse Event after completing Period 1.) | 8
Completed | 8 | 7 | 8
Not Completed | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | TAK-648 Sequence ABC | TAK-648 Sequence BCA | TAK-648 Sequence CAB
Started | 8 | 7 | 7 (1 Participant was withdrawn due to an Adverse Event after completing Period 2.)
Completed | 8 | 7 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set included of all participants who were enrolled and received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | TAK-648 Sequence ABC | TAK-648 Sequence BCA | TAK-648 Sequence CAB | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (8.26) | 35.3 (11.00) | 34.4 (9.91) | 33.7 (9.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 2 | 9
  Male | 6 | 3 | 6 | 15
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 4 | 6 | 3 | 13
  Not Hispanic or Latino | 4 | 2 | 5 | 11
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 1 | 2 | 0 | 3
  White | 6 | 6 | 8 | 20
  Multiracial | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 24
Height [Mean (Standard Deviation); unit: cm] | 175.6 (13.22) | 163.4 (11.07) | 171.4 (4.98) | 170.1 (11.18)
Weight [Mean (Standard Deviation); unit: kg] | 77.46 (18.762) | 70.11 (9.447) | 81.41 (7.596) | 76.33 (13.219)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.76 (2.350) | 26.24 (2.349) | 27.68 (1.709) | 26.23 (2.393)

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-648
Time Frame: Day 1 pre-dose and multiple timepoints post-dose (Up to 72 hours) in each Period
Population: The PK Set included all participants who received at least 1 dose of study drug and had at least 1 measurable postdose plasma concentration.
Measure: Mean (Standard Deviation); unit: mg/mL
Groups:
- TAK-648 Regimen A: TAK-648 0.3 mg, tablet, orally, 30 minutes after a high fat meal, once on Day 1 of Period 1, 2 or 3.
- TAK-648 Regimen B: Regimen B TAK-648 0.3 mg, tablet, orally, in fasted state, once on Day 1 of Period 1, 2 or 3.
- TAK-648 Regimen C: Regimen C TAK-648 0.3 mg, solution, orally, in fasted state, once on Day 1 of Period 1, 2 or 3.
Arm/Group | TAK-648 Regimen A | TAK-648 Regimen B | TAK-648 Regimen C
Number analyzed (Participants) | 23 | 23 | 23
mg/mL | 4.504 (1.2363) | 4.707 (1.5255) | 5.185 (1.9749)
Statistical Analysis 1: Comparison: TAK-648 Regimen A vs TAK-648 Regimen B; Test type: Superiority or Other; Point Estimate = 0.9660, 90% CI 2-sided [0.8747 to 1.0668] — Relative Bioavailability A/B. The point estimates and 90% CIs were obtained from the exponentiated results of the analysis of the natural logarithm-transformed data
Statistical Analysis 2: Comparison: TAK-648 Regimen B vs TAK-648 Regimen C; Test type: Superiority or Other; Point Estimate = 0.9223, 90% CI 2-sided [0.8352 to 1.0185] — Relative Bioavailability B/C. The point estimates and 90% CIs were obtained from the exponentiated results of the analysis of the natural logarithm-transformed data

2. Primary Outcome: AUClast: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-648
Time Frame: Day 1 pre-dose and multiple timepoints post-dose (Up to 72 hours) in each Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | TAK-648 Regimen A | TAK-648 Regimen B | TAK-648 Regimen C
Number analyzed (Participants) | 23 | 23 | 23
ng*hr/mL | 34.855 (8.8481) | 34.526 (9.2767) | 34.916 (10.7221)
Statistical Analysis 1: Comparison: TAK-648 Regimen A vs TAK-648 Regimen B; Test type: Superiority or Other; Point Estimate = 0.9998, 90% CI 2-sided [0.9540 to 1.0477] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: TAK-648 Regimen B vs TAK-648 Regimen C; Test type: Superiority or Other; Point Estimate = 1.0149, 90% CI 2-sided [0.9685 to 1.0636] — [estimate comment as in outcome 1, analysis 2]

3. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-648
Time Frame: Day 1 pre-dose and multiple timepoints post-dose (Up to 72 hours) in each Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | TAK-648 Regimen A | TAK-648 Regimen B | TAK-648 Regimen C
Number analyzed (Participants) | 23 | 23 | 23
ng*hr/mL | 35.241 (8.9283) | 34.922 (9.3106) | 35.353 (10.7619)
Statistical Analysis 1: Comparison: TAK-648 Regimen A vs TAK-648 Regimen B; Test type: Superiority or Other; Point Estimate = 0.9992, 90% CI 2-sided [0.9541 to 1.0464] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: TAK-648 Regimen B vs TAK-648 Regimen C; Test type: Superiority or Other; Point Estimate = 1.0134, 90% CI 2-sided [0.9676 to 1.0612] — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: Percentage of Participants Who Experience at Least One Treatment Emergent Adverse Event (TEAE)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: First dose of study drug to 30 days after the last dose of study drug (Up to Day 47)
Population: Safety Set included of all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | TAK-648 Regimen A | TAK-648 Regimen B | TAK-648 Regimen C
Number analyzed (Participants) | 23 | 23 | 23
percentage of participants | 17.4 | 8.7 | 0.0

5. Secondary Outcome: Percentage of Participants With Markedly Abnormal Laboratory Values at Least Once Post-dose
Time Frame: First dose of study drug to 7 days after the last dose of study drug (Up to Day 24)
Population: Safety Set included of all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | TAK-648 Regimen A | TAK-648 Regimen B | TAK-648 Regimen C
Number analyzed (Participants) | 23 | 23 | 23
percentage of participants | 4.3 | 4.3 | 0

6. Secondary Outcome: Percentage of Participants With Markedly Abnormal Vital Sign Values at Least Once Post-dose
Description: Vital signs included body temperature (oral), sitting blood pressure (after 5 minutes resting), respiration rate and pulse (beats per minute [bpm]).
Time Frame: First dose of study drug to 7 days after the last dose of study drug (Up to Day 24)
Population: Safety Set included of all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | TAK-648 Regimen A | TAK-648 Regimen B | TAK-648 Regimen C
Number analyzed (Participants) | 23 | 23 | 23
percentage of participants | 39.1 | 47.8 | 60.9

ADVERSE EVENTS:
Time Frame: First dose of study drug to 30 days after last dose (Up to Day 47)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TAK-648 Regimen A | TAK-648 Regimen B | TAK-648 Regimen C
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 4/23 | 2/23 | 0/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-648 Regimen A (N=23) | TAK-648 Regimen B (N=23) | TAK-648 Regimen C (N=23)
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Heart rate irregular (Investigations) | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.